CLINICAL TRIAL: NCT03194659
Title: Maternal Choline Supplementation and Its Impact on Docosahexaenoic Acid Supply in Human Pregnancy
Brief Title: Synergy Between Choline and DHA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cornell University (Other)
Collaborators: Balchem Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB #: 1702006936
Record Dates: First submitted 2017-06-13; First posted 2017-06-21 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Pregnancy
Keywords: Nutrition; choline; pregnancy; docosahexaenoic acid; DHA; fatty acids
MeSH Terms: interventions — Choline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All investigators interacting with participants will be masked to the study arm assignment. Only the Primary Investigator and Laboratory Manager (prepares supplements) will have access to participant's study assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (No Intervention): Administration of the deuterated choline chloride will take place in a grape juice cocktail solution. For individuals in the placebo arm of the trial, no additional choline chloride will be added to the cocktail.
- Supplemental Choline (Experimental): Administration of the deuterated choline chloride will take place in a grape juice cocktail solution. For individuals in the experimental arm of the trial, supplemental choline chloride will be added to the cocktail.
  Interventions: Dietary Supplement: Choline

INTERVENTIONS:
Dietary Supplement: Choline — Choline chloride is a water soluble choline salt that will be provided in a juice solution to participants to be consumed daily. The intervention will increase dietary choline intake by 500mg/day.
  Arms: Supplemental Choline

SUMMARY:
The purpose of this study is to determine whether choline supplementation influences the availability of docosahexaenoic acid throughout pregnancy.

DETAILED DESCRIPTION:
Metabolic synergy exists between choline, phospholipid, and polyunsaturated fatty acid metabolism. Previous evidence from our laboratory has shown that higher dietary choline intakes increase the amount of docosahexaenoic acid (DHA) incorporated into phosphatidylcholine (PC), as measured by PC-DHA concentrations in circulating erythrocytes. PC-DHA results from the production of PC through the phosphatidyl N-ethanolamine methyltransferase (PEMT) pathway and is critical for exporting fat from the liver to peripheral tissues. We are expanding this work to pregnant women, for whom DHA intake is critical to support the developing infant's growth, by undertaking a double blind, randomized controlled trial of choline supplementation (500mg) throughout the 2nd and 3rd trimesters of pregnancy. All women will consume 200mg of docosahexaenoic acid (DHA), a prenatal vitamin, and 25-50mg of deuterated choline (choline d9) daily throughout the duration of the trial. The use of a stable isotope will allow for modeling of choline dynamics throughout the 2nd and 3rd trimester of pregnancy, and calculate the activity of PEMT in pregnant women. Consenting participants will provide a baseline blood draw, followed by 2 additional blood draws throughout their pregnancies, and maternal/cord blood at birth, in addition to the placenta. This trial will test the hypothesis that choline supplementation increases the amount of PC-DHA in the blood of pregnant women and increase its supply to the developing fetus.

ELIGIBILITY:
Inclusion Criteria:

* healthy, singleton pregnant women gestational weeks 12-16, ages 21-40, willingness to comply with the study protocol

Exclusion Criteria:

* Habitually high choline/DHA intake
* Pre-pregnancy BMI >32
* Pregnancy complications and comorbidities (at baseline and throughout the study)
* Current smokers, drinkers, or drug users

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2017-10-05 (Actual); Primary Completion 2021-12-05 (Estimated); Study Completion 2021-12-05 (Estimated)

PRIMARY OUTCOMES:
DHA-Containing Phosphatidylcholine Species in Circulating Erythrocytes | Gestational Weeks 12-16 through Gestational Weeks 38-41
  Phosphatidylcholine species contain 2 fatty acid tails; phosphatidylcholines containing DHA at either the sn-1 or sn-2 positions are found circulating in erythrocytes and serve as a long term marker of DHA status. Erythrocyte PC-DHA is partially supplied by albumin bound lysophosphatidylcholine enriched with DHA, a product of the phosphatidylethanolamine methyltransferase pathway in the liver, which has been shown to be sensitive to dietary choline intakes in non-pregnant women.

SECONDARY OUTCOMES:
Circulating labeled and unlabeled choline metabolites in maternal plasma | Gestational Weeks 12-16 through Gestational Weeks 38-41
  The concentrations and isotopic enrichments of choline and its metabolites (betaine, dimethylglycine,sarcosine, total phosphatidylcholine) will be determined in the maternal, placental and fetal compartments by Liquid Chromatography Tandem Mass Spectrometry
The impact of dietary choline on total DHA concentrations in the maternal, fetal and placental compartments | Gestational Weeks 12-16 through Gestational Weeks 38-41
  The total concentrations of docosahexaenoic acid (DHA; % total fatty acids as determined by Gas Chromatography-Flame Ionization Detector) will be measured in the maternal blood throughout this study. Additionally, at term, placenta and cord blood will be collected and analyzed for total DHA measurements.
The Association of Maternal Choline Supplementation with Infant Visual Recognition Memory Novelty Score | 5, 7, 10, and 13 months of age
  The composite novelty score (proportion of looking to the novel image) is obtained from a series of 9 visual paired comparison tests. The novelty score is a measure of visual recognition memory for infants and has been shown to predict cognitive outcomes in childhood.
The Association of Maternal Choline Supplementation with Infant Visual Attention Orienting Speed Score | 5, 7, 10, and 13 months of age
  Visual attention orienting speed is measured by the latency to initiate a stimulus-guided fixation shift to a peripheral visual target (mean of up to 20 target presentations). The orienting score was found to be sensitive to maternal choline supplementation in infants of this age and has shown acceptable test-retest reliability and prediction of attention, memory, and intelligence quotient outcomes in childhood.
The Association of Maternal Choline Supplementation with Infant Sustained Focused Attention Score | 5, 7, 10, and 13 months of age
  Sustained focused attention is measured during a 5-minute period in which infants are engaged in solitary play with a complex toy. The score is the average duration of infant engagement in a state of focused attention on the toy. Infants who sustain focused attention for longer durations have been found to have fewer attentional problems as children.
The Association of Maternal Choline Supplementation with Infant Recall Memory Score | 13 months of age
  Recall memory is measured with a deferred imitation protocol. The infant watches an adult perform a novel sequence of actions on a set of objects to produce an interesting result. After a distraction-filled 15-minute delay the infant is given the objects and encouraged to engage in the modeled actions. The score is the number of target actions reproduced (average of 3 problems). Infants who achieve greater recall memory scores perform better on tests of memory during childhood.

OTHER OUTCOMES:
Maternal choline intake and microbiome composition | Gestational Weeks 12-16 through Gestational Weeks 38-41 and neonatal month 3
  Assess the effect of maternal choline intake during pregnancy on the maternal and neonatal gut microbiome, and the effect of the maternal microbiome on biomarkers of maternal status.

CONTACTS AND LOCATIONS:
Overall Officials: Marie A. Caudill, PhD, RD, Principal Investigator — Cornell University
Locations (1):
- Human Metabolic Research Unit, Cornell University, Ithaca, New York, United States

REFERENCES:
- [Derived] Klatt KC, McDougall MQ, Malysheva OV, Taesuwan S, Loinard-Gonzalez AAP, Nevins JEH, Beckman K, Bhawal R, Anderson E, Zhang S, Bender E, Jackson KH, King DJ, Dyer RA, Devapatla S, Vidavalur R, Brenna JT, Caudill MA. Prenatal choline supplementation improves biomarkers of maternal docosahexaenoic acid (DHA) status among pregnant participants consuming supplemental DHA: a randomized controlled trial. Am J Clin Nutr. 2022 Sep 2;116(3):820-832. doi: 10.1093/ajcn/nqac147. PMID 35575618